CLINICAL TRIAL: NCT04532775
Title: The Efficacy Of Magnesium In Radicular Lower Limb Pain When It Is Added To Local Anesthetics And Steroids In The Transforaminal Epidural Injections. A Comparative Study
Brief Title: Efficacy Of Magnesium In Radicular Pain When Added To Local Anesthetics And Steroids In Transforaminal Epidural Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, mohammed awad alsaeid ahmed, lecturer, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R139
Record Dates: First submitted 2020-08-20; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Neuropathy; Pain
Keywords: Magnesium; Transforaminal epidural; Steroids
MeSH Terms: conditions — Pain | interventions — Magnesium; Magnesium Sulfate; Methylprednisolone; Bupivacaine; Sodium Chloride; Isotonic Solutions

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled blinded study
Who Masked: Participant, Investigator
Masking Description: drugs used in this study are used within covered color coded syringes and participants are randomized to any of study groups via sealed opaque envelopes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group C (Other): This study was conducted on 100 patients. Patients were divided according to the injected drugs into two equal groups (50 patients each):
  1- Group (C): where all patients received through the transforaminal epidural approach 2 ml of bupivacaine (0.5%), 1ml of methylprednisolone (40 mg) and 1 ml of normal saline (0.9 %) with a total volume of 4 ml.
  Interventions: Drug: Methylprednisolone; Drug: Bupivacaine Hydrochloride; Drug: saline 0.9%
- group M (Other): 2- Group (M): where all patients received through the transforaminal epidural approach 2 ml of bupivacaine (0.5%), 1ml of methylprednisolone (40 mg) and 1 ml of preservative free magnesium (200 mg) with a total volume of 4 ml. Methylprednisolone which was used in this study was supplied from E.I.P.I.C.O pharmaceuticals -Egypt under license of UPJOHN s.a Puurs-Belgium (Depo-Medrol). Preservative free magnesium which was used in the study was prepared in McGuff Pharmaceuticals, Inc. Laboratories and supplied in 50 ml vials containing magnesium (200 mg/ml).
  Interventions: Drug: magnesium; Drug: Methylprednisolone; Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: magnesium — Preservative free magnesium which was used in the study was prepared in McGuff Pharmaceuticals, Inc. Laboratories and supplied in 50 ml vials containing magnesium (200 mg/ml).
  Other Names: magnesium sulphate
  Arms: group M
Drug: Methylprednisolone — Methylprednisolone which was used in this study was supplied from E.I.P.I.C.O pharmaceuticals -Egypt under license of UPJOHN s.a Puurs-Belgium (Depo-Medrol).
  Other Names: depomedrol
Drug: Bupivacaine Hydrochloride — local anesthetic drug
  Other Names: marcaine
Drug: saline 0.9% — solution for intravenous and epidural injection
  Other Names: isotonic solution
  Arms: group C

SUMMARY:
investigators want to assess the efficacy of magnesium in radicular lower limb pain when it is added to local anesthetics and steroids in the transforaminal epidural injections.

DETAILED DESCRIPTION:
INTRODUCTION:

One of the common presentation of low back pain and lower extremities pain is lumbar radicular pain which may be caused by a herniated intervertebral disc exerting a pressure on nerve roots, resulting in pain, functional disability, opioid use for pain relief and consuming health resources (1,2). Radicular pain has a typical shocking, lancinating, or electric character traveling into the lower limb along a narrow band. In approximately 90% of cases, radiculopathy is mainly due to a prolapsed disc causing nerve root impingement (3). Different modalities of treatments are used in managing chronic low back pain and radiculopathy. Most of the patients will respond well to conservative management. But after the failure of this conservative treatment, either surgical or nonsurgical modalities such as epidural injections are going to be considered in the treatment of lumbar radiculopathy (4). Transforaminal epidural injection (TFEI) is a known approach for treatment of spinal nerve root pathology. A transforaminal epidural directs medications at the nerve root as it leaves the spinal cord at the ventrolateral aspect of the epidural space whereas a conventional (interlaminar) epidural results in a small amount of medication over a wide area at the posterior epidural space (5). A transforaminal epidural gives us the opportunity to allocate the medications where they are required (6). Transforaminal epidural injections under fluoroscopic guidance have emerged as the preferred approach to the epidural space (7). Many drugs have been proven to be effective in managing low back pain when they are injected in the epidural space by transforaminal approach such as local anesthetics, steroids and adjuvants (7). Magnesium is a physiological blocker of the NMDA receptors (8) because it blocks NMDA channels in a voltage-dependent manner, and such NMDA antagonist effect can inhibit the induction of central sensitization from peripheral nociceptive stimulation (9,10). Magnesium may suppress neuropathic pain (11), enhance morphine analgesia, attenuate morphine tolerance (12), and improve fentanyl analgesia when magnesium is given intrathecally (13). Magnesium deficiency produces hyperalgesia (14) and has been related to cause some acute medical and surgical conditions in which pain or stress is present (15). Magnesium is proved to be injected safely within the nervous tissue in animals (16) and in 2002 Asokumar and his colleagues proved that magnesium is safely injected Intrathecal in human (17). Because of the results of a previous study that indicates that intrathecal administration of sulfate sault in magnesium has a risk of neurotoxicity (18), investigators preferred to use preservative free magnesium in our study. The aim of this study was to evaluate the efficacy of magnesium sulphate as an anti-neuropathic drug in relieving unilateral lower limb radicular pain due to disc prolapse when it was injected with lidocaine and steroids in the anterior epidural space using the transforaminal epidural approach. Our primary outcome was to assess the improvement of pain score post-injection, while, the secondary outcome was to evaluate the improvement of the functional ability and the satisfaction level of the patients after the procedure.

Patients and Methods:

Firstly, The study IS approved by the local ethics committee (Fayoum Faculty of Medicine Research Ethics Committee R139 ). This prospective, controlled, randomized, double-blinded study is going to be carried out in the pain management department of Fayoum University Hospital. Written consents are going to be taken from all patients. The randomization is going to be performed via sealed opaque envelopes. All procedures are going to be performed by one investigator who is blind to the injected drugs used in this study. Inclusion criteria are patients of both gender, aged from 20 up to 70 years old, American Society of Anesthesiologists (ASA) physical status grade I and II (19), admitted for pain management of their unilateral lower limb radicular pain due to lumbo-sacral disc prolapse confirmed by lumbo-sacral magnetic resonance imaging ( MRI) after failure of conservative treatments in the form of drug therapy and physiotherapy to control the pain for 6 weeks. Exclusion criteria are patients with axial back pain without leg radiation, patients with motor neurological deficits, previous spine surgeries, allergy to the study drugs used, uncontrolled diabetes mellitus or hypertension, local or systemic infection, pregnancy, and patients with any other neurological deficits as cauda equina. This study is going to be conducted on 100 patients. Patients are going to be divided according to the injected drugs into two equal groups (50 patients each):

1. Group (C): where all patients will receive through the transforaminal epidural approach 2 ml of bupivacaine (0.5%), 1ml of methylprednisolone (40 mg) and 1 ml of normal saline (0.9 %) with a total volume of 4 ml.
2. Group (M): where all patients will receive through the transforaminal epidural approach 2 ml of bupivacaine (0.5%), 1ml of methylprednisolone (40 mg) and 1 ml of preservative free magnesium (200 mg) with a total volume of 4 ml. Methylprednisolone which is used in this study is going to be supplied from E.I.P.I.C.O pharmaceuticals -Egypt under license of UPJOHN s.a Puurs-Belgium (Depo-Medrol). Preservative free magnesium which is used in the study is prepared in McGuff Pharmaceuticals, Inc. Laboratories and supplied in 50 ml vials containing magnesium (200 mg/ml).

All patients are going to be evaluated pre-operatively by medical history, clinical examination, and lumbosacral spine MRI. The severity of pain is going to be assessed using the visual analog scale (VAS) where 0 and 10 were marked on a 10cm linear scale (0- 4 mm = no pain, 5-44 mm = mild pain, 45- 74 = moderate pain, 75-100 = severe pain) (20). Patients are going to be evaluated for effective pain relief (defined as ≥50% reduction of pain perception post-intervention by VAS. Functional assessment is done using Modified Oswestry Disability Questionnaire (MODQ), which is formed of a10 item scale with six response categories each. Each item scores from 0 to 5, higher scores being worse, which is transformed into a 0-100 scale. The ten items include pain intensity, personal care, lifting, walking, sitting, standing, sleeping, work, social life and traveling. Patients with scores between 0 to 20 have Minimal Disability, between 21 and 40 have Moderate Disability, between 41-60 have Severe Disability, 61 to 80 are crippled and 81 to 100 are bed-bound or exaggerating their symptoms, this questionnaire has been designed to give us information about how back or leg pain is affecting the ability to manage in everyday life (21). VAS and MODQ are going to be assessed immediately pre-intervention and at 1 day, 1 week, 1 month, and 3 months post-intervention.

The demographic data for all patients as regards to age, gender, weight, and height are going to be recorded and compared between the studied groups. Also, the pre-intervention clinical examination data of all patients as regards to the level, the site of disc prolapse, and the side of radiculopathy are going to be recorded and compared between the groups. The occurrence of side effects is going to be recorded and compared between both groups post-intervention.

The level of the intervention (affected nerve root) and the right versus the left sides of radiating pain are going to be determined by both clinical examination and radiological findings. Pre-intervention, an intravenous (IV) cannula is going to be inserted with initiation of normal saline (0.9%) at a rate of 10 ml/kg to prevent hypotension. Emergency drugs as atropine and ephedrine are going to be prepared. All patients are going to be monitored throughout the procedure by electrocardiogram (ECG), noninvasive blood pressure, and pulse oximetry throughout the procedure and during the post-interventional time for 2 hours. Patients are going to be placed in a prone position with a pillow under their abdomen (between the iliac crests) to decrease the lumbar lordosis. Mild sedation is going to be given with 0.02 mg/kg of midazolam intravenously. TFEIs are going to be done under full sterile technique using fluoroscopic guidance. After fluoroscopic detection of the desired intervertebral level, the entry site is identified, and the skin is anesthetized with local infiltration of 3 ml of lidocaine 1%. TFEI approach is performed under biplane fluoroscopic guidance. While a patient lying in the prone position, the tube is rotated obliquely approximately 10-30° toward the affected side to ensure injection at the neural foramen. The goal of positioning is to allow a perpendicular needle tract toward the classic injection site below the pedicle (22).

Sample size calculation:

The required sample size has been calculated using the G*Power version 3.1.9 Software (Faul et al., 2007) (23). The primary outcome measure is the proportion of patients achieving satisfactory response at 12 weeks after the procedure. Satisfactory response is defined as reduction of the pain score by 50% or more from the pre-procedure value. Since no previous study has compared the effect of adding magnesium sulfate or steroid to local anesthetic for transforaminal block in patients with chronic LBP, investigators considered that a medium effect size corresponding to a Cohen's ω of 0.3 would be clinically relevant. So, investigators calculated that a sample size of 44 patients in either study group would achieve a power of 80% to detect statistical significance for an effect size equivalent to Cohen's ω of 0.3 regarding the proportion of patients achieving satisfactory response at 12 week after the procedure using a two-sided chi-squared test with an alpha error of 0.05. Considering a drop-out rate of around 10%, 50 patients will be recruited in either group.

ELIGIBILITY:
Inclusion criteria were:

* Patients of both gender.
* Patients aged from 20 up to 70 years old.
* Patients of American Society of Anesthesiologists (ASA) physical status grade I and II.
* Patients admitted for pain management of their unilateral lower limb radicular pain due to lumbo-sacral disc prolapse confirmed by lumbo-sacral magnetic resonance imaging ( MRI) after failure of conservative treatments in the form of drug therapy and physiotherapy to control the pain for 6 weeks.

Exclusion criteria were:

* Patients with axial back pain without leg radiation.
* Patients with motor neurological deficits.
* Previous spine surgeries.
* Allergy to the study drugs used.
* Uncontrolled diabetes mellitus or hypertension.
* Local or systemic infection.
* Pregnancy.
* Patients with any other neurological deficits as cauda equina.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-30 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is going to be assessing the improvement of pain score post-injection | 3 monthes
  The severity of pain was assessed using the visual analog scale (VAS) where 0 and 10 were marked on a 10cm linear scale (0- 4 mm = no pain, 5-44 mm = mild pain, 45- 74 = moderate pain, 75-100 = severe pain) (20). Patients were evaluated for effective pain relief (defined as ≥50% reduction of pain perception post-intervention by VAS

SECONDARY OUTCOMES:
the secondary outcome is going to be evaluating the improvement of the functional ability of the patients after the procedure | 3 monthes
  Functional assessment was done using Modified Oswestry Disability Questionnaire (MODQ), which is formed of a10 item scale with six response categories each. Each item scores from 0 to 5, higher scores being worse, which is transformed into a 0-100 scale. The ten items include pain intensity, personal care, lifting, walking, sitting, standing, sleeping, work, social life and traveling. Patients with scores between 0 to 20 have Minimal Disability, between 21 and 40 have Moderate Disability, between 41-60 have Severe Disability, 61 to 80 are crippled and 81 to 100 are bed-bound or exaggerating their symptoms, this questionnaire has been designed to give us information about how back or leg pain is affecting the ability to manage in everyday life.
age | preinjection
  in years
weight | preinjection
  kilograms
gender | preinjection
  male and female
height | preinjection
  centimetres
level of disc prolapse | preinjection
  lumbar or sacral levels
side of disc prolapse | preinjection
  right or left
site of disc prolapse | preinjection
  central, paracentral or lateral

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Awad M, Raouf MM, Mikhail HK, Megalla SA, Hamawy TY, Mohamed AH. Efficacy of transforaminal epidural magnesium administration when combined with a local anaesthetic and steroid in the management of lower limb radicular pain. Eur J Pain. 2021 Jul;25(6):1274-1282. doi: 10.1002/ejp.1748. Epub 2021 Mar 16. PMID 33559245